CLINICAL TRIAL: NCT05351502
Title: A Phase 1, Open-Label, Dose Escalation and Dose Expansion Study to Assess the Safety and Efficacy of Nitric Oxide Injection Into Unresectable Solid Cutaneous/Subcutaneous Primary or Metastatic Tumors
Brief Title: A Study to Assess the Safety and Efficacy of Nitric Oxide Injection Into Unresectable Solid Primary or Metastatic Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beyond Air Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BA-ONC-01
Record Dates: First submitted 2022-04-12; First posted 2022-04-28 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-07

CONDITIONS: Cancer
Keywords: Intratumoral Injection; Nitric Oxide; single gNO injection
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: In Part A, the following gNO doses will be studied to determine MTD and/or OBD: 25,000 ppm, 50,000 ppm and 100,000 ppm. Additional dose levels may be evaluated based on the emerging data as determined by the Safety Review Committee.
  Once the MTD and/or OBD is determined, additional patients will be treated in Part B Dose Expansion to further characterize the safety and biomarkers of gNO and determine RP2D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): Subjects will receive 25,000 ppm NO
  Interventions: Drug: Nitric Oxide 25,000 ppm
- Cohort 2 (Experimental): Subjects will receive 50,000 ppm NO
  Interventions: Drug: Nitric Oxide 50,000 ppm
- Cohort 3 (Experimental): Subjects will receive 100,000 ppm NO
  Interventions: Drug: Nitric Oxide 100,000 ppm
- RP2D Expansion (Experimental): Subjects will receive the RP2D dose of NO
  Interventions: Drug: Nitric Oxide selected dose

INTERVENTIONS:
Drug: Nitric Oxide 25,000 ppm — Intratumoral injection of 25,000 gNO
  Other Names: gNO injection
  Arms: Cohort 1
Drug: Nitric Oxide 50,000 ppm — Intratumoral injection of 50000 gNO
  Arms: Cohort 2
Drug: Nitric Oxide 100,000 ppm — Intratumoral injection of 100,000 gNO
  Arms: Cohort 3
Drug: Nitric Oxide selected dose — Intratumoral injection of selected does on gNO
  Arms: RP2D Expansion

SUMMARY:
This is a Phase 1, open-label, dose-escalation and dose-expansion study comprised of a screening period, a single treatment session, an evaluation period of 21±3 days, and safety and survival follow-up period of up to 12 weeks post-treatment.

DETAILED DESCRIPTION:
The purpose of this Phase 1 study is to initiate clinical development of gNO in patients with unresectable cutaneous or subcutaneous primary or metastatic solid tumors that are not amenable or have failed standard treatment, for which no therapy of proven efficacy exists, or which has progressed despite standard therapy. This study of gNO treatment will consist of 2 parts: a dose-escalation part to establish a safe and tolerable dose of gNO in patients with primary or metastatic unresectable cutaneous or subcutaneous solid tumors (Part A), and a dose expansion phase (Part B) which may be initiated at the Sponsor's discretion after the maximum tolerated dose (MTD) and/or optimal biological dose (OBD) (or recommended Phase 2 dose [RP2D]) has been determined in the dose-escalation phase (Part A). This study will be the basis for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient (male or female) is at least 18 years of age at the time of signature of the informed consent form.
* Patient has an ECOG Performance Status score of 0-3 and with a life expectancy of ≥3 months.
* Patient must have a confirmed diagnosis of at least one unresectable cutaneous or subcutaneous histologically confirmed primary or metastatic solid tumor. Up to five target lesions may be identified.
* No therapy of proven efficacy exists for the tumor, the tumor is not amenable to standard therapies, the tumor has failed to respond to standard therapy or has progressed despite standard therapy.
* Patient has measurable disease on imaging based on RECIST Version 1.1.
* Patient have adequate hematologic and organ function.
* Patient have not had radiotherapy to the targeted lesions within the preceding 12 months.
* Superficial tumor axis minimum length and depth of 4.5mm. .
* Patient is not with childbearing potential or agrees to use adequate contraceptive methods

Exclusion Criteria:

* The tumor is situated in the lymph node, in thyroid, close to trachea or in facial area or other region which, in the Investigator's opinion, can pose extra risk to the patient.
* Has received prior systemic anti-cancer therapy including investigational agents within 14 days of the start of study treatment.
* Active central nervous system tumors or metastases..
* Received systemic corticosteroid therapy ≤1 week prior to study treatment or any other form of systemic immunosuppressive medication for medically significant acute or chronic conditions.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, neuropathy and protocol-defined laboratory values.
* Active or prior documented autoimmune or inflammatory disorders.
* History of primary immunodeficiency, history of allogenic organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of enrolment.
* Known active infection and uncontrolled intercurrent illness.
* Receiving drugs that have contraindication with NO.
* Patient is receiving anticoagulants including low molecular weight heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-08-14 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs, SAEs and DLTs (safety) parameters. | up to12 weeks from injection
  The incidence and characteristics of adverse events (AEs), serious adverse events (SAEs), dose-limiting toxicities (DLTs) and changes in assessed safety parameters. Toxicity will be graded according to NCI CTCAE version 5.0

SECONDARY OUTCOMES:
Anti-tumor activity of a single intratumoral gNO injection at all administered doses | up to Day 21 from injection
  The anti-tumor activity of a single intratumoral gNO injection will be measured per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, and secondarily immune-related RECIST (iRECIST).

OTHER OUTCOMES:
Assessment of predictive biomarkers for anti-tumor activity of a single intratumoral gNO injection | up to Day 21 from injection
  Measurement of blood immune biomarkers levels

CONTACTS AND LOCATIONS:
Overall Officials: David Greenberg, MD, Study Director — Study Internal Medical Monitor
Locations (4):
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Hadassah Ein-Karem, Jerusalem
  - Sheba Medical Center, Ramat Ef‘al
  - Sourasky Tel Aviv Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Meirovitz A., et al. Phase 1 study of ultra-high concentration nitric oxide (UNO) in relapsed or refractory, unresectable, primary, or metastatic cutaneous and subcutaneous malignancies. SITC 2023 — https://jitc.bmj.com/content/11/Suppl_1/A827
- See also: Confino H., et al. Intratumoral administration of high-concentration nitric oxide and anti PD-1 treatment leads to higher tumor regression rates and prolonged survival in CT26 tumor-bearing mice SITC 2022 — https://jitc.bmj.com/content/10/Suppl_2/A855